CLINICAL TRIAL: NCT04545372
Title: Effect of Aerobic Exercises on Immune System in Patients With Multiple Sclerosis
Brief Title: Aerobic Exercises for Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Nehad Ahmed Youness Abo-zaid, Lecturer of physical therapy, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/001072
Record Dates: First submitted 2020-08-26; First posted 2020-09-11 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Multiple Sclerosis, Primary Progressive
Keywords: Multiple Sclerosis; Aerobic exercises; cytokine IL-10; cytokine IL-17
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: study group (GA) and control group (GB) in addition to normal matched subjects (GC).The control group (GB)was treated by the disease modifying drug (interferon beta-1a) "Rebif", (GA) treated by the same drug in addition to a physical therapy program of aerobic exercises for 40 min included bicycle ergometry training
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator) Single (Outcomes Assessor) Blinding process to participants and care providers was impossible due to the nature of intervention therapy. Data were analyzed by an impartial statistician (outcomes assessor), referring to each arm with an encoded name: Group A (study group) and Group B (control group),
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the study group (Experimental): the study group (GA) was treated only by the disease modifying drug (interferon beta-1a) in addition to aerobic exercise.
  Interventions: Other: aerobic exercise
- the control group (No Intervention): control group (GB)was treated only by the disease modifying drug (interferon beta-1a)

INTERVENTIONS:
Other: aerobic exercise
  Arms: the study group

SUMMARY:
Multiple sclerosis (MS) is a chronic inflammatory demyelinating disease of the central nervous system (CNS) .It is the most common neurological disorders affecting young adults.Multiple sclerosis is an autoimmune disease that results in progressive neural degeneration. Cytokines play an important role in the pathogenesis and treatment of MS.

DETAILED DESCRIPTION:
This research aims to evaluate the effect of aerobic exercises on the immune system anti-inflammatory (IL-10) and pro inflammatory (IL-17) cytokines and its consequences on the functional status in the Multiple Sclerosis patients.

Aerobic exercises are a term to describe planned, structured and repetitive physical activity undertaken over a prolonged period to maintain or improve physical fitness and functional capacity .

ELIGIBILITY:
Inclusion Criteria:

age ranged from 25 to 45 years. All the patients were remitting relapsing MS according to (revised McDonald criteria.

Duration of MS disease was one to two years before starting of the study. Last attack occurred three months ago. All patients were able to ambulate

Exclusion Criteria:

Patients with other neurological deficits , patient with significant orthopedic abnormalities for both lower limbs, patient with contracture , patient with deformities, pregnant females

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-02-02 (Actual); Primary Completion 2018-08-04 (Actual); Study Completion 2020-08-06 (Actual)

PRIMARY OUTCOMES:
blood analysis | serum anti inflammatory cytokine IL-10, will be assessed at 0 day
  serum anti inflammatory cytokine IL-10,
blood analysis | serum anti inflammatory cytokine IL-10, wil lbe assessed at 90 day
  serum anti inflammatory cytokine IL-10,
blood analysis | pro inflammatory cytokine IL-17 will be assessed at 0 day
  pro inflammatory cytokine IL-17
blood analysis | pro inflammatory cytokine IL-17 will be assessed at 90 day
  pro inflammatory cytokine IL-17

CONTACTS AND LOCATIONS:
Overall Officials: Nehad A. Abo-Zaid, Ph.D, Principal Investigator — South Valley University; Heba A. Kalifa, Ph.D, Principal Investigator — Cairo University
Locations (1):
- South Valley University, Faculty of Physical Therapy, Qina, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Steensberg A, Fischer CP, Keller C, Moller K, Pedersen BK. IL-6 enhances plasma IL-1ra, IL-10, and cortisol in humans. Am J Physiol Endocrinol Metab. 2003 Aug;285(2):E433-7. doi: 10.1152/ajpendo.00074.2003. PMID 12857678
- [Background] Barry A, Cronin O, Ryan AM, Sweeney B, Yap SM, O'Toole O, Allen AP, Clarke G, O'Halloran KD, Downer EJ. Impact of Exercise on Innate Immunity in Multiple Sclerosis Progression and Symptomatology. Front Physiol. 2016 Jun 2;7:194. doi: 10.3389/fphys.2016.00194. eCollection 2016. PMID 27313534
- [Background] Haegert DG. Multiple sclerosis: a disorder of altered T-cell homeostasis. Mult Scler Int. 2011;2011:461304. doi: 10.1155/2011/461304. Epub 2011 Sep 15. PMID 22096637
- [Background] Broughton SE, Hercus TR, Lopez AF, Parker MW. Cytokine receptor activation at the cell surface. Curr Opin Struct Biol. 2012 Jun;22(3):350-9. doi: 10.1016/j.sbi.2012.03.015. Epub 2012 Apr 20. PMID 22521507
- [Background] McDonald WI, Compston A, Edan G, Goodkin D, Hartung HP, Lublin FD, McFarland HF, Paty DW, Polman CH, Reingold SC, Sandberg-Wollheim M, Sibley W, Thompson A, van den Noort S, Weinshenker BY, Wolinsky JS. Recommended diagnostic criteria for multiple sclerosis: guidelines from the International Panel on the diagnosis of multiple sclerosis. Ann Neurol. 2001 Jul;50(1):121-7. doi: 10.1002/ana.1032. PMID 11456302

DOCUMENTS (1):
  • Study Protocol (2020-08-30): https://cdn.clinicaltrials.gov/large-docs/72/NCT04545372/Prot_000.pdf